CLINICAL TRIAL: NCT02562495
Title: Interest of the Ultrasound to Evaluate the Quadriceps Muscle Wasting in Critical Ill Patients.
Brief Title: Ultrasound to Evaluate the Quadriceps Muscle Wasting
Acronym: ECHOSCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1508123; 2015-A01204-45 (Other: ANSM)
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Severe Cerebral Pathology
Keywords: severe cerebral pathology; Ultrasound; thickness of the quadriceps
MeSH Terms: interventions — Tomography, X-Ray Computed; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT scan and Ultrasonography (Experimental): Up to three measurements (CT scan and Ultrasonography), will be made concurrently between the day of admission (D1) in intensive care unit and the tenth day ( D10 ) .
  Interventions: Device: CT Scan and ultrasonography

INTERVENTIONS:
Device: CT Scan and ultrasonography — Up to three measurements (CT scan and Ultrasonography) of the thickness of quadriceps, will be made concurrently .

SUMMARY:
Intensive care unit acquired muscle weakness (ICUAW) is a common disease. After 7 days of mechanical ventilation, a quarter of patients develop an ICUAW responsible of a 15-20% of muscle loss. This is a serious pathology associated with high morbidity and mortality.

Clinical diagnosis of ICUAW is difficult and need a patient awoken. CT scan and Magnetic Resonance Imaging (MRI) are considered as "gold standards" to quantify and monitor changes in muscle mass. But these tools are not adapted to ICU patients.

Ultrasound (US) is an easy access tool at the bedside to assess muscle mass and does not expose the patient to additional radiation.

The objective of this study is to evaluate the correlation between US and CT scan to measure quadriceps muscle thickness of ICU patients.

DETAILED DESCRIPTION:
As part of the monitoring of the neurological disease, brain CT scans are frequently performed. At the same time, an acquisition sequence centered on the quadriceps will follow the brain sequences. Up to three brain CT scans coupled with a quadriceps imaging will be performed between the day of admission and on the tenth day of hospitalization. An ultrasound of the quadriceps will be performed concomitantly. The thickness of the quadriceps is measured by an independent operator on CT and ultrasound images.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years admitted to intensive care for a severe brain injury (Glasgow <8) and with a predictive duration of mechanical of at least 48hours

Exclusion Criteria:

* Pregnancy,
* Bilateral trauma of thighs,
* Coma induced by poisoning or by a metabolic disorder,
* Morbid obesity (BMI > 35).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Concordance of the measurement of the quadriceps thickness by ultrasound and by CT scan | Between the day of admission (D1) in intensive care unit and the tenth day ( D10 )
  Concordance of each of the three measurements of the thickness of quadriceps realised concurrently by CT scan and Ultrasonography (composite measure)

SECONDARY OUTCOMES:
kinetic of the thickness of quadriceps | Between the day of admission (D1) in intensive care unit and the tenth day ( D10 )
  Evolution of he thickness of quadriceps measure concurrently by CT scan and Ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme MOREL, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No